CLINICAL TRIAL: NCT02297802
Title: A Phase I Single Patient IND for PD-0325901
Brief Title: A Single Patient IND for PD-0325901
Status: No longer available | Type: Expanded Access
Sponsor: Sharp HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: 130596 SHRP
Record Dates: First submitted 2014-05-12; First posted 2014-11-21 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Prior Treatment With PD-0325901 With Ongoing Clinical Response
MeSH Terms: interventions — mirdametinib

INTERVENTIONS:
Drug: PD-0325901

SUMMARY:
The purpose of this study is to provide access for a single patient to PD-0325901 who was previously enrolled in a phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Prior treatment with PD-0325901 with ongoing response

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Healthcare, San Diego, California, United States